CLINICAL TRIAL: NCT05567237
Title: Effects of Microcurrent Treatment With and Without Resistance Exercises on Body Composition, Muscle Strength, and Physical Function in Middle-aged Adults
Brief Title: Effects of Microcurrent Treatment With and Without Resistance Exercises
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Greenwich (Other)
Responsible Party: Principal Investigator, Fernando Naclerio, Professor, University of Greenwich
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HUS0120
Record Dates: First submitted 2022-09-12; First posted 2022-10-05 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Sarcopenia; Ageing Well
Keywords: microcurrent; resistance exercises; adults; MENS
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind parallel-group between-participants design, which will analyse the effects of microcurrent on health-related parameters. Once considered eligible, the participants will be randomly assigned to the following two groups:
  1. Microcurrent (MC)
  2. Sham (SH) Thereafter, all of the participants will be offered to take part in a supervised resistance training (RT) programme which will be combined with either the MC or SH intervention.
  The participants who do not accept to undergo the resistance training programme will integrate a non-exercise group involving a 6-week intervention period using the microcurrent (MC) or the sham (SH) device. Those participants who accept to perform the resistance training programme (regardless of being previously allocated to MC + RT or SH + RT) will perform a 2-session familiarization before the beginning of the study. Then, they will follow the exercise programme of 2 training sessions per week for 6 weeks (12 sessions in all).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a randomised, balanced, double-blind parallel-group between-participants design. The participants will not know whether they receive sham or live microcurrent. Both devices (microcurrent and sham) will look exactly the same in terms of appearance, colour, size and weight. The current transmitted from the microcurrent device is insufficient to stimulate sensory nerve fibres, so participants will not be able to feel it, and due to the fact that the devices will have the same appearance, neither participants nor researchers will be able to identify those participants allocated to the MC or the SH groups. Only one researcher who will not be involved in the assessments and training supervision will know the participant allocation during the intervention (unblinded researcher).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Microcurrent alone (MC) (Active Comparator): This group will receive a live microcurrent device and they will not be engaged in any resistance training exercises.
  Interventions: Other: Microcurrent treatment
- Microcurrent with exercise (MC + RT) (Active Comparator): This group will receive a live microcurrent device and they will follow an exercise programme of 2 training sessions per week for 6 weeks (12 sessions in all)
  Interventions: Other: Microcurrent treatment with resistance exercise programme
- Sham alone (SH) (Sham Comparator): This group will receive a sham microcurrent device and they will not be engaged in any resistance training exercises.
  Interventions: Other: No treatment
- Sham with exercise (SH + RT) (Sham Comparator): This group will receive a sham microcurrent device and they will follow an exercise programme of 2 training sessions per week for 6 weeks (12 sessions in all)
  Interventions: Other: Resistance exercise programme

INTERVENTIONS:
Other: Microcurrent treatment with resistance exercise programme — This intervention will allow us to explore the effects of microcurrent added to resistance exercise.
  Arms: Microcurrent with exercise (MC + RT)
Other: Resistance exercise programme — This intervention works as a control group for the participants undergoing the exercise programme.
  Arms: Sham with exercise (SH + RT)
Other: Microcurrent treatment — This intervention will allow us to explore the effects of microcurrent alone.
  Arms: Microcurrent alone (MC)
Other: No treatment — This intervention works as a control group for the participants who are not taking part into the exercise programme.
  Arms: Sham alone (SH)

SUMMARY:
* Aim: to analyse the effects of microcurrent treatment alone, and combined with a resistance exercise programme, on muscle strength, body composition and physical functional capacity in middle-aged adults.
* Methods

  * Randomised, balanced, double-blind parallel-group between-participants design.
  * Participants - non-regularly trained adults (people who do not engage regularly in physical sessions), aged 40 to 65 years old.
  * All participants will be invited to take part in a 6-week supervised resistance training programme that will be combined with microcurrent (MC) or sham (SH) intervention. The participants who do not accept to undergo the resistance training programme will integrate a non-exercise group involving a 6-week intervention period using the microcurrent (MC) or the sham (SH) device. The devices will be provided by Arc4Health (ARC Microtech Ltd, UK; https://arcmicrotech.com/arc4health/). The device Arc4Health has regulatory approval as a Class IIa medical device in the areas of pain management and tissue repair.

The following will be analysed:

1. Microcurrent alone (MC)
2. Microcurrent with exercise (MC + RT)
3. Sham alone (SH)
4. Sham with exercise (SH + RT)

   * The participants who agree to take part in the training programme will have 2 sessions a week for a period of 6 weeks. The training programme involves elastic bands and is designed to increase strength and muscle mass.
   * Measurements of body composition (via plethysmography BodPod), strength, functional capacity, muscular structure (via non-invasive ultrasound), and immunological blood markers will be undertaken at baseline and after the 6-week intervention period.

DETAILED DESCRIPTION:
Microcurrent therapy is non-invasive method that provides different frequencies and transmits tiny currents through the skin within the range of milliamperes (<1 mA). Human studies demonstrated that microcurrent can reduce the severity of symptoms of muscle damage induced by exercise protocols in healthy men, healthy men and women, trained men, and cross-country male athletes. To the best of the authors' knowledge, no formal research has been conducted to verify the effects of microcurrent added to resistance exercises on physical function in non-trained middle-aged adults. Therefore, it is important to understand to what extent the application of microcurrent added to physical exercises (the hallmark of prevention and treatment of sarcopenia) can slow the age-related decline of muscular function and play a role in the prevention of sarcopenia.

Aim: To analyse the effects of microcurrent treatment alone, and combined with a resistance exercise programme, on muscle strength, body composition and physical function in middle-aged adults.

Hypotheses (i) Microcurrent alone will counteract the loss of muscle mass and strength which accompanies ageing, and it will improve functional capacity and wellbeing compared to a sham, non-microcurrent treatment, in individuals with a low level of physical activity (sedentary population who are not engaged in regular exercise programmes).

(ii) The application of microcurrent alone, although not improving strength, will counteract the loss of muscle mass and strength in sedentary individuals.

(iii) Adding a resistance training programme to microcurrent treatment will optimise exercise-induced outcomes, allowing superior gains in muscle mass, strength, functional capacity, and wellbeing, compared to the application of microcurrent alone.

Experimental design

The study involves a 6-week randomised, balanced, double-blind parallel group between-participants design, which will analyse the effects of microcurrent on health-related parameters. Once considered eligible, the participants will be randomly assigned to the following two groups:

1. Microcurrent (MC)
2. Sham (SH) All participants will be offered to take part in a supervised resistance training (RT) programme which will be combined with either the MC or SH intervention.

The participants who do not accept to undergo the resistance training programme will integrate a non-exercise group involving a 6-week intervention period using the microcurrent (MC) or the sham (SH) device. Those participants who accept to perform the resistance training programme (regardless of being previously allocated to MC + RT or SH + RT) will perform a 2-session familiarization before the beginning of the study. Then, they will follow the exercise programme of 2 training sessions per week for 6 weeks (12 sessions in all).

Participants will wear the microcurrent or sham device on the dominant upper arm for a period of 3 hours every day. For those included in the exercise group, the device will be used immediately after each training session, and in the mornings on the non-training days. For those included in the non-exercise group, the device will be worn in the mornings. Measurements of body composition, muscle thickness, functional capacity, and blood indices of health and wellbeing will be determined before (T1) and after the 6-week intervention period (T2).

In summary, the following four treatment conditions are expected to be analysed:

(i) Microcurrent alone (MC) (ii) Microcurrent with exercise (MC + RT) (iii) Sham alone (SH) (iv) Sham with exercise (SH + RT)

Intervention Familiarization period The participants from the MC+RT and SH+RT groups will undertake 2 sessions (on 2 non-consecutive days in 1 week) of familiarization, supervised by a qualified strength and conditioning instructor (graduate or MSc student). The familiarization aims to instruct the participants on how to perform the selected exercises, control breathing and control intensity. The Rate of Perceived Exertion OMNI-RES scale will be used to control the level of resistance and monitor participants' progression. The proposed OMNI-RES scale with elastic bands was previously validated for prescribing exercise intensity with TheraBand resistance bands in older adults.

During the familiarization, participants will be asked to execute 1 set of 10 reps with different resistance bands (and with different grip widths) to establish the initial level of resistance, which will be thereafter scheduled for the intervention. The elastic bands will be marked with numerical points 3 cm apart throughout the band to objectify the grip width. A few attempts of each exercise will be allowed in order to find, and objectively feel the correct resistance. Once the resistance level is achieved, the colour and the corresponding bandwidth will be recorded for each participant in each particular exercise.

Resistance Training Programme (RT) The RT programme will be performed over a 6-week (12 sessions in total) training intervention using elastic bands.

The RT programme involves 8 multi-joint and single-joint exercises targeting the whole-body musculature. The exercises will be performed in the following order: 1. Squat with shoulder press, 2. Biceps curl, 3. Squat, 4. Lat-pull down, 5. Deadlift, 6. Triceps extension, 7. Lunge, and 8. Upright row. The participants will perform 3 sets of 12 to 15 repetitions with ~1.5 to 2 min rest between sets of each exercise. The estimated duration of each workout is 60 min including a standardised 10-min warm-up with dynamic and static flexibility exercises (10 min).

The participants will be surveyed to find out whether middle-aged and older people prefer to perform the exercise programme (RT) in a group supervised face-to-face setting at our Avery Hill Campus, or in their home following a pre-recorded video session or live session. The current COVID restrictions on physical activities which take place in venues will also be considered. It will be anticipated that all sessions are conducted under the supervision (live or online) of at least one qualified instructor on non-consecutive days (48 hours apart). To avoid dropout of participants, giving them the opportunity to train at their convenient time by watching a pre-recorded RT online session (and submitting a short google form immediately after completing the workout online) will also be considered.

Training load

As indicated earlier, the participants will execute 3 sets of a minimum of 12 to a maximum of 15 repetitions of each exercise with ~1.5 to 2 min rest between sets (consisting of stretching elements without the use of the bands). The following progression model protocol will be implemented:

* First block (week 1) - participants should reach a rate of perceived exertion (RPE) of 6 to a maximum of 7 at the end of each set of 12 reps. When an RPE lower than 6 is reported at the end of the set, the participant will be asked to increase the number of repetitions to a maximum of 15 in the subsequent sets, always maintaining a final RPE no higher than 7.
* Second block (week 2) - participants should reach an RPE of 7 to a maximum of 8 at the end of each set of 12 reps. When an RPE lower than 7 is reported at the end of the set, the participant will be asked to increase the number of repetitions to a maximum of 15 in the subsequent sets, always maintaining a final RPE no higher than 8.
* Third block (week 3 to week 6) - participants should reach an RPE of 8 to a maximum of 9 at the end of each set of 12 reps. When an RPE lower than 8 is reported at the end of the set, the participant will be asked to increase the number of repetitions to a maximum of 15 in the subsequent sets, always maintaining a final RPE no higher than 9. For those participants who still feel that the effort is easier than the expected rate, the magnitude of the resistance can be increased by shortening the grip width of the band or changing to a different band colour/level offering a higher resistance.

Intervention protocol (microcurrent or sham device) The Arc4Health microcurrent device (approved as a Class IIa medical device in the areas of pain management and tissue repair) will be used in the study.

Participants will wear the microcurrent or sham device on the dominant upper arm for 3 hours every day (after each session on a training day and in the morning on all other days) or in every morning for those who are not taking part in the resistance training. It is expected that participants will be exposed to 21 hours of microcurrent (Programme 1) or sham stimulus per week (a total of 126 hrs for 6 weeks).

Expected outcomes from the investigation It is expected that results from the current project will demonstrate the potential benefits of microcurrent treatment alone and combine microcurrent with resistance training to maximise the benefits on body composition, muscle strength, and muscle function in middle-aged adults.

ELIGIBILITY:
Inclusion Criteria:

* non-regularly trained male and female adults, aged 40 to 65 years old.

Exclusion Criteria:

* with no musculoskeletal injuries, metabolic conditions, or diseases or currently taking medications, smoking, and nutritional supplements known to affect physical performance, muscle damage or recovery processes (e.g., creatine, whey protein, and amino acids, vitamin, or mineral supplementation, etc.) within 6 weeks prior to the start of the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Change of body fat | The body fat will be assessed to measure changes at week 6.
  Air displacement plethysmography (BodPod) will be used to calculate the percentage of body fat of the participants. Measurements will be collected in kg and then the percentage relative to body mass will be calculated.
Change of muscle thickness | The muscle thickness will be measured to track changes at week 6.
  Using Ultrasound (Affiniti 50 Ultrasound system) to measure thickness of Elbow flexors (Brachialis and Biceps) and Vastus Lateralis. Measurements will be collected in millimeters

SECONDARY OUTCOMES:
Changes Neutrophils to Lymphocyte ratio (NLR) | The white blood cells count will be measured to track changes at week 6.
  White blood cells will be measured by using the HemoCue® WBC DIFF System. Values of Neutrophils to Lymphocytes will be collected in 10(9)/L

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Naclerio, PhD, Principal Investigator — University of Greenwich
Locations (1):
- School of Human Sciences, University of Greenwich, Avery Hill Campus, Sparrows Farm, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available

REFERENCES:
- [Background] Naclerio F, Moreno-Perez D, Seijo M, Karsten B, Larrosa M, Garcia-Merino JAL, Thirkell J, Larumbe-Zabala E. Effects of adding post-workout microcurrent in males cross country athletes. Eur J Sport Sci. 2021 Dec;21(12):1708-1717. doi: 10.1080/17461391.2020.1862305. Epub 2021 Feb 8. PMID 33295832
- [Background] Naclerio F, Seijo M, Karsten B, Brooker G, Carbone L, Thirkell J, Larumbe-Zabala E. Effectiveness of combining microcurrent with resistance training in trained males. Eur J Appl Physiol. 2019 Dec;119(11-12):2641-2653. doi: 10.1007/s00421-019-04243-1. Epub 2019 Oct 17. PMID 31624949